CLINICAL TRIAL: NCT03200262
Title: Analytic and Functional Evaluation After Surgical Treatment Using an Original Arthroscopic Trillat Technique in Patients With Chronic Anterior Shoulder Instability
Acronym: TRILLARTHRO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: ORTA 2016 bis
Record Dates: First submitted 2017-06-21; First posted 2017-06-27 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Chronic Anterior Shoulder Instability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The shoulder is the most mobile joint in the body, and the most exposed to the risk of dislocation notably anterior. Chronic instability of the shoulder is frequent after dislocation, and principally affects people who are young and active. It can have major functional repercussions, leading to restricted participation in professional or sports activities, even in everyday life activities.

Surgical stabilisation is the reference treatment for chronic anterior shoulder instability, and has given good results. There are numerous surgical techniques available; the orthopaedists at Dijon CHU now practice the Bristow-Trillat technique under arthroscopy, following many years of reflexion and adaptation.

Rehabilitation following the surgery is essential, notably to recover muscle strength in the shoulder rotator cuff after surgery, which correlates directly with dynamic stability of the joint. At the moment, we do not know the objective evolution of muscle strength after the Trillat arthroscopic technique.

The isokinetic evaluation of muscle strength in the rotator cuff has been validated and is reproducible. It gives objective and reliable values for muscle strength, thus making it possible to guide and to optimise rehabilitation protocols done by patients under the supervision of a physiotherapist, and to estimate time to the return to physical, professional or sports activities, without risk.

ELIGIBILITY:
Inclusion Criteria:

* Persons informed about the research
* Male or female
* Age between 16 and 45 years
* Regular sport activity (leisure or competition)
* First surgical indication for stabilisation using the Trillat arthroscopic technique
* Patient operated on using the Trillat arthroscopic technique for chronic anterior shoulder instability in the orthopaedic and trauma unit of Dijon CHU

Exclusion Criteria:

* Persons without health insurance cover
* Concomitant, disabling shoulder joint disease inflammatory rheumatism, which could be exacerbated by the tests
* Associated lesions in the shoulder: rupture of rotator cuff tendons, neurological lesions, bone lesions: fracture of the neck of humerus, of the greater tubercle or the coracoid process
* Paraplegia and peripheral neurological disease
* Surgery other than the Trillat arthroscopic technique alone
* Treatment with the Trillat arthroscopic technique as second line, after failure of the first strategy
* Contralateral history of dislocation with surgical repair
* History of disease with excess laxity (collagen disease, Marfan, Elhers-Danlos)
* History of debilitating pain in the back, elbows or wrists
* Contra-indication for isokinetic tests
* Cognitive disorders
* Major post-operative complications delaying the rehabilitation
* Early recurrence of dislocation after surgery
* Post-operative immobilisation protocol not respected

Ages: 16 Years to 45 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients with chronic anterior shoulder instability treated with surgery using an original Trillat arthroscopic technique
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from maximum muscle torque in patients who have undergone surgical treatment for chronic anterior shoulder instability before and after surgery using the Trillat arthroscopic technique | Baseline, 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France